CLINICAL TRIAL: NCT03589313
Title: Evaluation of the Pharmacokinetics, Safety and Tolerability of a Single Dose of GLPG3067 Administered as Solid Formulation in Male Subjects With Cystic Fibrosis.
Brief Title: Pharmacokinetics of GLPG3067 in Male Subjects With Cystic Fibrosis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLPG3067-CL-104; 2017-002294-19 (EudraCT Number)
Record Dates: First submitted 2018-07-09; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLPG3067 single dose. (Experimental): Single Dose of GLPG3067 film coated tablets.
  Interventions: Drug: GLPG3067 single dose

INTERVENTIONS:
Drug: GLPG3067 single dose — GLPG3067 film coated tablets provided at Day 1.

SUMMARY:
This clinical study is a Phase I, open-label, single-center study designed to evaluate the pharmacokinetics profile of a single oral dose of GLPG3067 in adult male subjects with cystic fibrosis in fed state.

ELIGIBILITY:
Inclusion Criteria:

* Male subject ≥18 years of age on the day of signing the ICF.
* A confirmed clinical diagnosis of CF.
* Exocrine pancreatic insufficiency (documented in the subject's medical record).
* Stable concomitant medication regimen for pulmonary health for at least 2 weeks prior to study drug administration

Exclusion Criteria:

* History of clinically meaningful unstable or uncontrolled chronic disease that makes the subject unsuitable for inclusion in the study in the opinion of the investigator.
* Unstable pulmonary status or respiratory tract infection (including rhinosinusitis) requiring a change in therapy within 2 weeks prior to study drug administration.
* Need for supplemental oxygen during the day, and >2 L/minute while sleeping.
* History of solid organ or hematopoietic cell transplantation.
* History of hepatic cirrhosis with portal hypertension (e.g., signs/symptoms of splenomegaly, esophageal varices).
* Use of CFTR modulator therapy (e.g., lumacaftor or ivacaftor) within 2 weeks prior to study drug administration.
* Abnormal liver function test at screening, defined as aspartate aminotransferase (AST) and/or ALT and/or alkaline phosphatase and/or gamma-glutamyl transferase (GGT) ≥3x the upper limit of normal, and/or total bilirubin ≥1.5x the upper limit of normal.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (cmax) of GLPG3067 single dose. | Between Day 1 pre-dose and Day 4.
  To evaluate the PK profile of GLPG3067 after a single oral dose of GLPG3067.
Area under the plasma concentration-time curve from time zero until 24 hours post-dose ( (AUC0-24h) of GLPG3067 single dose. | Between Day 1 pre-dose and Day 4.
  To evaluate the PK profile of GLPG3067 after a single oral dose of GLPG3067.
Area under the plasma concentration-time curve from time zero until 72 hours post-dose (AUC0-72h) of GLPG3067 single dose. | Between Day 1 pre-dose and Day 4.
  To evaluate the PK profile of GLPG3067 after a single oral dose of GLPG3067.

SECONDARY OUTCOMES:
The number of subjects with adverse events. | From screening to 19 days after the last dose.
  To evaluate the safety and tolerability of a single oral dose of GLPG3067 in adult male subjects with CF.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Van de Steen, MD MBA, Study Director — Galapagos NV
Locations (1):
- University Hospital Leuven,Pediatric Pulmonology, Leuven, Belgium